CLINICAL TRIAL: NCT07299539
Title: Impact on Mortality of the Choice Between a Mono- Versus Combination Antibiotic Therapy in Enterococcus Faecalis Bacteremia
Brief Title: Treatment of Enterococcus Faecalis Bacterem
Acronym: E-faecalis
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9378
Record Dates: First submitted 2025-12-09; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Enterococcus Faecalis Bacteremia
Keywords: Enterococcus faecalis bacteremia; Mortality; Monotherapy versus combination therapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Enterococcus faecalis is a germ frequently responsible for bacteremia which can be severe with 15-25% risk of mortality and 26% risk of infectious endocarditis. There is no recommendation for the treatment of "simple" Enterococcus faecalis bacteremia (meaning without infectious endocarditis at diagnosis), nor studies comparing monotherapy versus combination antibiotic therapy.

Our main objective is to study the impact on mortality of bacteriostatic monotherapy and bactericidal combination antibiotic therapy in patients with Enterococcus faecalis bacteremia. We aim to also study the mortality up to three months, the failures of treatment, the modalities of treatment, the renal toxicity and the bacterial resistance.

ELIGIBILITY:
Inclusion Criteria:

* Subject of legal age (≥18 years)
* Having a positive blood culture result for Enterococcus faecalis identified within the microbiology laboratory of the University Hospital of Strasbourg during the period from 01 January 2017 to 31 December 2023.

Exclusion Criteria:

* Penicillin treatment < 7 days
* Treatment not containing a penicillin effective against enterococci among those studied: amoxicillin or piperacillin-tazobactam
* Combination of penicillin with another antibiotic effective against enterococci other than cephalosporins or aminoglycosides (glycopeptides, linezolids, carbapenems, levofloxacin, moxifloxacin).
* Bacteremia with one or more other pathogens within the first 7 days of bacteremia
* Infective endocarditis at diagnosis and within the first 7 effective days of treatment
* Resistance of Enterococcus faecalis to amoxicillin
* Mortality <72 hours after initiation of antibiotic therapy
* Lack of information regarding the chosen antibiotic treatment

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult subject having a positive blood culture result for Enterococcus faecalis identified within the microbiology laboratory of the University Hospital of Strasbourg during the period from 01 January 2017 to 31 December 2023.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2024-02-24 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Intrahospital all-cause mortality | Up to 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Service des Maladies Infectieuses et Tropicales - CHU de Strasbourg - France, Strasbourg, France